# **Statistical Analysis Plan**

| Protocol Title: | A Phase 2b Dose Ranging Study to Evaluate the Efficacy and Safety of Efavaleukin Alfa in Subjects with Active Systemic Lupus Erythematosus With Inadequate Response to Standard of Care Therapy (VIOLET) | |
|---|---|---|
| Short Protocol Title: | Efficacy and Safety of Efav with Active Systemic Lupus | - |
| Protocol Number: | 20200234 | |
| NCT Number: | NCT04680637 | |
| Authors: | | |
| Sponsor: | Amgen Inc. One Amgen Center Drive, Thousand Oaks, CA 91320 | , USA |
| SAP Date: | <u>Document Version</u> | <u>Date</u> |
| | Original (v1.0) | 26 October 2021 |
| | Amendment 1 | 29 November 2022 |
| | Amendment 2 | 25 September 2023 |

| Version Number | Date (DDMMMYYYY) | Summary of Changes, including rationale for changes |
|---|---|---|
| Original (v1.0) | 26OCT2021 | |
| Amendment 1 | 29NOV2022 | Incorporate changes in protocol amendment 3: |



Product: Efavaleukin Alfa Protocol Number: 20200234 Date: 25 September 2023


| Amendment 2 | 25SEP2023 | Administrative, typographical and formatting changes throughout. Incorporate changes in the scope of planned analyses due to early termination of the study: |
|---|---|---|
| | | <ul> <li>Removed subsequent IAs following study early termination</li> <li>Removed some exploratory endpoints</li> <li>Removed statistical comparisons of treatment groups; descriptive statistics by treatment groups will be generated instead</li> </ul> |

# **Table of Contents**

| Tab | le of C | ontents | 3 |
|-----|---------|------------------------------------------------|----|
| 1. | Intro | duction | 8 |
| 2. | Obje | ctives, Endpoints and Hypotheses | 8 |
| | 2.1 | Objectives and Endpoints/Estimands | |
| | 2.2 | Hypotheses and/or Estimations | |
| 3. | Stud | y Overview | 11 |
| | 3.1 | Study Design | 11 |
| | 3.2 | Sample Size | 13 |
| | 3.3 | Adaptive Design | |
| 4. | Cova | ariates and Subgroups | 15 |
| | 4.1 | Planned Covariates | |
| | 4.2 | Subgroups | 15 |
| 5. | Defir | nitions | 15 |
| | 5.1 | Basic Definition | 15 |
| | 5.2 | Study Points of Reference | 17 |
| | 5.3 | Study Dates | |
| | 5.4 | Study Time Intervals | |
| | 5.5 | Arithmetic Calculations | 18 |
| | 5.6 | Efficacy Assessments | 19 |
| | 5.7 | Patient-reported Outcome (PRO) Assessments | 24 |
| 6. | Analy | ysis Sets | 26 |
| | 6.1 | Full Analysis Set | 26 |
| | 6.2 | Safety Analysis Set | 26 |
| | 6.3 | Interim Analyses Set(s) | 26 |
| 7. | Plani | ned Analyses | 26 |
| | 7.1 | Interim Analysis and Early Stopping Guidelines | 26 |
| | 7.2 | Final Analysis | 28 |
| 8. | Data | Screening and Acceptance | 29 |
| | 8.1 | General Principles | 29 |
| | 8.2 | Data Handling and Electronic Transfer of Data | |
| | 8.3 | Handling of Missing and Incomplete Data | |
| | 8.4 | Detection of Bias | |
| | 8.5 | Outliers | |
| | 8.6 | Distributional Characteristics | |
| | 8.7 | Validation of Statistical Analyses | 32 |
| 9. | Statis | stical Methods of Analysis | 33 |



| | 9.1 | Genera | al Considerations | 33 |
|---|---|---|---|---|
| | 9.2 | Subject | t Accountability | 33 |
| | 9.3 | Importa | ant Protocol Deviations | 33 |
| | 9.4 | Demog | raphic and Baseline Characteristics | 33 |
| | 9.5 | Efficacy | y Analyses | 36 |
| | 9.6 | Safety | Analyses | 39 |
| | | 9.6.1 | Adverse Events | 39 |
| | | 9.6.2 | Laboratory Test Results | 40 |
| | | 9.6.3 | Vital Signs | 40 |
| | | 9.6.4 | Electrocardiogram | 40 |
| | | 9.6.6 | Exposure to Investigational Product | 41 |
| | | 9.6.7 | Exposure to Other Protocol-permitted Therapy | 41 |
| | | 9.6.8 | Exposure to Concomitant Medication | 41 |
| | 9.7 | Other A | Analyses | 41 |
| | | 9.7.1 | Analyses of Pharmacokinetic Endpoints | 41 |
| | | 9.7.2 | Analyses of Clinical Outcome Assessments | 42 |
| | | 9.7.3 | Analyses of Biomarker Endpoints | 42 |
| 10. | Chan | ges From | Protocol-specified Analyses | 42 |
| 11. | Litera | iture Citat | tions / References | 42 |
| 12. | Appe | ndices | | 44 |
| | Appe | ndix A. F | Reference Values/Toxicity Grades | 44 |
| | Appe | ndix B. S | SLE Assessment Forms/Instruments | 45 |
| | | | Patient-reported Outcome Forms/Instruments | |
| | | | Analytical Windows | |
| | Appe | ndix E. H | landling of Dates, Incomplete Dates and Missing Dates | 64 |



# **List of Tables**

| Table 3-1 Analyses Schedule | 16 |
|--------------------------------------------------------|----|
| Table 9-1. Primary Efficacy Endpoint Summary Table | 40 |
| Table 9-2. Secondary Efficacy Endpoint Summary Table | 42 |
| Table 9-3. Exploratory Efficacy Endpoint Summary Table | 44 |
| Table 9-4 Selected Safety Laboratory Tests | 51 |

# **List of Figures**

No table of figures entries found.



# **List of Abbreviations**

| Abbreviation | Explanation |
|---|---|
| ACR | American College of Rheumatology |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| ANCOVA | analysis of covariance |
| Anti-dsDNA | anti-double stranded DNA |
| AST | aspartate aminotransferase |
| ВНМ | Bayesian Hierarchical Model |
| BICLA | BILAG based Combined Lupus Assessment |
| BILAG | British Isles Lupus Assessment Group |
| CLASI | Cutaneous Lupus Erythematosus Area and Severity Index |
| Clinical SLEDAI-2K | SLEDAI-2K assessment score without the inclusion of points attributable to any urine or laboratory results including immunologic parameters. |
| CNS | central nervous system |
| COVID-19 | Coronavirus Disease 2019 |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DMC | data monitoring committee |
| ECG | electrocardiogram |
| eCRF | Electronic Case Report Form |
| EOS | end of study |
| ET | early termination |
| FAS | Full Analysis Set |
| GLM | Generalized linear model |
| hSLEDAI | Hybrid Systemic Lupus Erythematosus Disease Activity Index |
| IA | interim analysis |
| IBG | Independent Biostatistics Group |
| Ig | immunoglobulin |
| IL-2 | interleukin 2 |
| IP | Investigational product |



| IPD | Important protocol deviation |
|-----------|----------------------------------------------------------|
| IRT | interactive response technology |
| LLDAS | Lupus Low Disease Activity State |
| NSAID | non-steroidal anti-inflammatory drugs |
| ocs | oral corticosteroids |
| PD | pharmacodynamic |
| PGA | Physician Global Assessment |
| PK | pharmacokinetic |
| PROMIS | Patient-Reported Outcome Measurement Information System |
| Q2W | every 2 weeks |
| RAR | Response Adaptive Randomization |
| SAP | statistical analysis plan |
| SF36v2 | Medical Outcomes Short Form 36 version 2 questionnaire |
| SLE | systemic lupus erythematosus |
| SLEDAI-2K | Systemic Lupus Erythematosus Disease Activity Index 2000 |
| SLICC | Systemic Lupus International Collaborating Clinics |
| SOC | standard of care |
| SRI | Systemic Lupus Erythematosus Responder Index |
| Treg | regulatory T cells |
| VAS | visual analog scale |



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


# 1. Introduction

**Objectives** 

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within the protocol amendment **3** for study 20200234, Efavaleukin Alfa dated **21 October 2022**. The scope of this plan **is reduced from those outlined in the protocol due to determination of futility at a preplanned interim analysis and subsequent study early termination. It includes the final analysis that is planned and will be executed by the Amgen Global Biostatistical Science department unless otherwise specified.** 

**Endpoints** 

# 2. Objectives, Endpoints and Hypotheses

# 2.1 Objectives and Endpoints/Estimands

| Objectives | Litapolita |
|---|---|
| Primary | |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa at week 52, as<br/>measured by the SRI-4 response</li> </ul> | SRI-4 response at week 52 |
| Primary Estimand | |
| <ul> <li>The primary estimand is the difference in SRI-4 response rates between each efavaleukin alfa dose group and placebo at week 52 for all subjects with SLE with inadequate response to SOC therapy who are randomized, regardless of investigational product compliance; subjects will be considered non-responders for using more than protocol-permitted therapies including:</li> <li>Subjects requiring a dose of systemic corticosteroids for SLE above their baseline dose after week 16</li> <li>Subjects requiring either dose increases of the current immunosuppressants/immunomodulators or initiation of new immunosuppressant/immunomodulator(s)</li> </ul> | |
| Secondary | |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa at week 52, as<br/>measured by the BICLA index<br/>responses</li> </ul> | BICLA response at week 52 |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa at week 52, as<br/>measured by LLDAS response</li> </ul> | LLDAS response at week 52 |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa at week 52, as<br/>measured by OCS tapering</li> </ul> | <ul> <li>Reduction of OCS to ≤ 7.5 mg/day<br/>by week 44 and sustained through<br/>week 52 in subjects with a<br/>baseline OCS dose ≥ 10 mg/day</li> </ul> |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa at week 24, as<br/>measured by SRI-4 response</li> </ul> | SRI-4 response at week 24 |



Product: Efavaleukin Alfa Protocol Number: 20200234 Date: 25 September 2023

| Evaluate the efficacy of<br>efavaleukin alfa at week 24, as<br>measured by the BICLA index<br>responses | BICLA response at week 24 |
|---|---|
| Evaluate the efficacy of efavaleukin alfa at weeks 24 and 52, as measured by hSLEDAI | <ul> <li>hSLEDAI response (i.e., reduction ≥ 4 points from baseline) at week 24</li> <li>hSLEDAI response (i.e., reduction</li> </ul> |
| | ≥ 4 points from baseline) at week 52 |
| Evaluate the efficacy of<br>efavaleukin alfa on joints and skin | <ul> <li>Improvement from baseline in tender and swollen joint count ≥ 50% at weeks 8, 12, 24, 36, and 52 in subjects with ≥ 6 tender and swollen joints involving hands and wrists at baseline</li> </ul> |
| | <ul> <li>Improvement from baseline in<br/>CLASI activity score ≥ 50% at<br/>week 8, 12, 24, 36, and 52 in<br/>subjects with a CLASI activity<br/>score ≥ 8 at baseline</li> </ul> |
| Evaluate the efficacy of<br>efavaleukin alfa using BILAG<br>score | <ul> <li>Annualized flare rate (as measured by BILAG score designation of "worse" or "new" resulting in a B score in ≥ 2 organs or an A score in ≥ 1 organ) over 52 weeks</li> </ul> |
| <ul> <li>Evaluate the efficacy of<br/>efavaleukin alfa using patient<br/>reported outcomes</li> </ul> | <ul> <li>Change from baseline in fatigue<br/>standardized score using the<br/>PROMIS Fatigue SF 7a at week<br/>12, 24, 36, and 52</li> </ul> |
| | <ul> <li>Change from baseline in the<br/>physical component score, mental<br/>component score and individual<br/>domains of the SF 36 v2 at week<br/>12, 24, 36, and 52</li> </ul> |
| | <ul> <li>Change from baseline in the<br/>domain scores on the Lupus QoL<br/>at weeks 12, 24, 36, and 52</li> </ul> |
| <ul> <li>Characterize the safety of<br/>efavaleukin alfa</li> </ul> | <ul> <li>Treatment-emergent adverse<br/>events</li> </ul> |
| | <ul> <li>Serious adverse events</li> </ul> |
| | <ul> <li>Clinically significant changes in<br/>laboratory values and vital signs</li> </ul> |



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


Characterize the PK of efavaleukin alfa
 Trough and sparse postdose serum concentrations of efavaleukin alfa

BICLA = British Isles Lupus Assessment Group Based Composite Lupus Assessment; CLASI = Cutaneous Lupus Erythematosus Area and Severity Index; hSLEDAI = Hybrid Systemic Lupus Erythematosus Disease Activity Index; IL-2 = interleukin-2; LLDAS = Lupus Low Disease Activity State; OCS = oral corticosteroid; PGA = Physician Global Assessment;

PK = pharmacokinetic(s); PROMIS Fatigue SF7A = Patient-Reported Outcome Measurement Information System Fatigue Short Form 7a Instrument; QoL = quality of life; SLE= systemic lupus erythematosus; SF36v2 = Medical Outcomes Short Form 36 version 2 Questionnaire; SOC = standard of care; SRI-4 = Systemic Lupus Erythematosus Responder Index;



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 



# 2.2 Hypotheses and/or Estimations

At least 1 efavaleukin alfa dose will have greater efficacy than placebo as measured by the SRI-4 response rate at week 52 in subjects with active SLE with inadequate response to SOC therapy who are randomized, regardless of investigational product compliance; subjects using more than protocol-permitted therapies will be considered as non-responders:

- Subjects requiring a dose of systemic corticosteroids for SLE above their baseline dose after week 16
- Subjects requiring either dose increases of the current immunosuppressants/immunomodulators or initiation of new immunosuppressant/immunomodulator(s).

# 3. Study Overview

#### 3.1 Study Design

This is a Bayesian adaptive phase 2b, multi-center, double-blind, randomized, placebo-controlled dose ranging study in subjects with active SLE and inadequate response to SOC therapies, including OCS, immunosuppressants, and immunomodulators. Previous biologic use is allowed with an adequate washout period.

The study design includes 3 active efavaleukin alfa treatment groups every 2 weeks [Q2W], Q2W, and Q2W) and a placebo group, SRI-4 response at week 52 as the primary endpoint, and an approximate sample size of 320 subjects.

Subjects will be randomized to receive either placebo or 1 of 3 doses of efavaleukin alfa for a duration of 52 weeks. The randomization ratio will start as 1:1:1:1, and then may be adapted at planned interim analyses (IAs) based on the clinical efficacy, as measured by SRI-4 response, using Response Adaptive Randomization (RAR) for the purpose of



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

allocating more subjects to more efficacious doses and fewer subjects to less efficacious doses, with a fixed 25% of subjects allocated to placebo throughout the study. The RAR will be implemented with a computerized system that assigns a treatment to subjects without unblinding any study personnel or Amgen study team members, including the investigators or subjects, to the subject's randomized treatment assignment or the current allocation ratio.

Study duration for a single subject will be 56 weeks (including the safety follow-up period) plus the screening period. Treatment will be administered every 2 weeks with the final dose at week 50. All subjects will be followed for safety for 6 weeks after the last dose of investigational product.

Subjects will undergo a screening visit to confirm eligibility requirements. At day 1 (baseline), prior to randomization, disease activity (clinical hybrid SLEDAI score  $\geq$  4) and stability and compliance of OCS and other immunosuppressant/immunomodulator doses, must be present. The maximum time between screening and randomization is 33 days. Subjects who do not meet all the eligibility requirements prior to randomization on day 1 will be considered screen failures. Subjects may be allowed to rescreen three times.

Immunosuppressant/immunomodulator dose(s) should remain stable through week 52. For OCS, initiation or temporary increases in OCS are allowed between weeks 0 to 10, provided that return to baseline dose occurs within the subsequent 2 weeks. OCS may be tapered after week 12 at the investigator's discretion but should not be changed during the last 8 weeks (week 44 to 52) of the 52-week treatment period.

Subjects who meet the criteria listed below will be allowed to continue the study but will be considered as experiencing treatment failure for the primary efficacy endpoint analyses:

- Subjects requiring a dose of systemic corticosteroids for SLE above their baseline dose after week 16
- Subjects requiring either dose increases of the current immunosuppressants/ immunomodulators or initiation of new immunosuppressant/ immunomodulator(s)

IAs will be conducted to allow for adaption of the randomization ratio for newly enrolled subjects to the 3 efavaleukin alfa treatment groups, holding the allocation to placebo



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

constant at 25%, and assessing efficacy for early futility or administrative success decisions:

 The study team, investigators, and subjects will remain blinded to the results of the IAs unless futility is determined.

- The first IA will be executed after the first 40 subjects are randomized and have had the opportunity to complete the week 24 assessment. Subsequent IAs are scheduled after every additional 32 subjects are randomized and have had the opportunity to complete the week 24 assessment until full enrollment or until futility is determined for all doses at an IA. The last IA will occur when all 320 subjects are randomized and have had the opportunity to complete the week 24 assessment. This IA will be referred to as the 'all-subjects-week-24 IA'. Analyses planned at each IA are listed in Table 3-1.
- Efficacy analyses will be performed at the IAs to assess the likelihood of each efavaleukin alfa treatment group being superior to placebo by a clinically meaningful difference.
  - From the second IA until before the last IA, if this likelihood is unacceptably low for all dose levels, the trial is recommended to stop for futility.
  - At the 'all-subjects-week-24 IA', if this likelihood is sufficiently high with at least one efavaleukin alfa dose level, this IA will trigger an administrative success signal. This would not alter the ongoing or planned activities of this phase 2b study, but downstream planning for subsequent trials (e.g., a phase 3 study) may commence.
- of the results from the 3<sup>rd</sup> IA and subsequent decision by the Data Access Plan Team, the study was terminated due to futility and further enrollment in the study was stopped. Previously enrolled subjects were discontinued from IP and terminated the study after being followed for an additional 6 weeks following last dose of IP. The remaining planned IAs, including the 4<sup>th</sup> to the last IA ('all-subjects-week-24-IA') were not conducted.

# 3.2 Sample Size

The approximate sample size of 320 subjects is chosen to provide approximately 80% power to detect ≥ 25% absolute improvement for at least 1 efavaleukin alfa dose group



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

relative to placebo in the primary endpoint of SRI-4 response rate at week 52 at a significance level of 0.025 (1-sided) using a Bayesian Hierarchical Model, assuming a 40% response rate in placebo group.

Because enrollment was stopped early, the actual sample size is smaller.

# 3.3 Adaptive Design

The prospectively defined adaptive features include RAR, early decision for futility and an early trigger for administrative success. The following adaptations are based on the planned IA results:

- Adaptive randomization begins after a fixed allocation period. After each IA (if before full enrolment), the randomization probability for each of the 3 active doses may be changed based on clinical efficacy after an IA, while the randomization allocation for placebo is kept constant at 25%.
- Efficacy is assessed against predefined early stopping rules for futility from the second IA until before the last IA. If futility is triggered, the study could be terminated, e.g., continued enrollment and IP dosing for previously enrolled subjects would be stopped, etc.
- Efficacy is assessed against predefined rules for early administrative success
  only at the last planned IA. If administrative success is determined, downstream
  activities may be planned/initiated, but the execution of the trial would not be
  stopped or altered.
- All adaptive decisions will be based on the SRI-4 response at week 52 with longitudinal modeling of SRI-4 response data. For a subject who has not yet completed through week 52, their 52-week value will be imputed using a longitudinal model based on their week 16, 20, or 24 SRI-4 response data, whichever is the latest.

Modeling and simulations were used to design this Bayesian adaptive trial and refine study design features to achieve optimal operating characteristics, including but not limited to type I error, power and estimation bias.

The IAs will be conducted by an Independent Biostatistics Group (IBG) and will be reviewed by a Data Monitoring Committee (DMC), both external to Amgen. The study team, investigators and subjects will remain blinded to the results of the IAs unless futility is determined.



Product: Efavaleukin Alfa Protocol Number: 20200234

Date: 25 September 2023 

**Table 3-1 Planned Analyses Schedule Decisions at Each Interim Analysis and Final Analysis** 

| Timepoint | Adaptive Decision | Number of subjects with opportunity to complete week 24 |
|---|---|---|
| 1 <sup>st</sup> IA | RAR | 40 |
| 2 <sup>nd</sup> IA | Futility, RAR | 72 |
| 3 <sup>rd</sup> IA | Futility, RAR | 104 |
| 4 <sup>th</sup> IA <sup>ac</sup> | Futility, RAR | 136 |
| 5 <sup>th</sup> IA <sup>ac</sup> | Futility, RAR | 168 |
| 6 <sup>th</sup> IA <sup>ac</sup> | Futility, RAR | 200 |
| 7 <sup>th</sup> IA <sup>ac</sup> | Futility, RAR | 232 |
| Last IA <sup>bc</sup> | Administrative success | 320 |
| Final Analysis | Not applicable | All subjects reach EOS |

IA = interim analysis; RAR = response adaptive randomization; EOS = end of study

#### 4. **Covariates and Subgroups**

#### 4.1 **Planned Covariates**

Not applicable.

#### 4.2 Subgroups

The primary endpoint will be **summarized** within each of the subgroups listed below. If the subgroup sample size is less than 10% of the population, this subgroup may not be evaluated. The subgroups of interest include the following:

- baseline hSLEDAI (< 10, ≥ 10)
- region (North America + Western Europe + Asia Pacific, ROW)

#### 5. **Definitions**

#### 5.1 **Basic Definition**

Investigational Product (IP)

Efavaleukin alfa and placebo.

**Enrollment/Randomization Date** 



<sup>&</sup>lt;sup>a</sup> Interim analyses are planned after every 32 subjects are randomized and have had the opportunity to complete the week 24 assessment until full enrollment or until futility is determined for all doses at an IA. Number of IAs will depend on the observed enrollment rate.

<sup>&</sup>lt;sup>b</sup> Last IA is the all-subjects-week-24 IA. The administrative success analysis at the last IA will not result in any adaptive decision for the ongoing study.

<sup>&</sup>lt;sup>c</sup> Canceled due to study early termination.

Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

The enrollment/randomization date is the date on which a subject is assigned to a treatment group by the IRT system.

#### **First Dose Date**

The first dose date is the date of administration of the first dose of IP; this may or may not be the same as randomization date.

#### **Actual Treatment Received**

The actual treatment received is the IP the subject actually received, regardless of what the subject was randomized to. In cases where a subject received both efavaleukin alfa and placebo, the actual treatment received will be the efavaleukin alfa dose. In cases where a subject received multiple different efavaleukin alfa doses, the actual treatment received will be based on the highest efavaleukin alfa dose received. In cases where the subject received more than efavaleukin alfa dose, the subject will be assigned to efavaleukin alfa dose.

# **Duration of IP exposure**

The duration of IP exposure will be derived as the date of the last IP administration plus 13 days (14-day window-1), end of study date or data cutoff date, whichever occurs first, minus the date of first IP administration plus 1 day.

#### Flare Exposure Time

The flare exposure time is the time from study day 1 up to the last flare assessment date.

# **Treatment-emergent adverse event**

Treatment-emergent adverse events are **defined as** events categorized as Adverse Events (AEs) starting on or after first dose of IP as determined by "Did event start before first dose of investigational product?" equal to "No" or missing on the Events eCRF and up to the end of study date.

#### **Baseline medication**

Baseline medication is defined as any medication with start date on or before study day 1 and ongoing while on study.

#### **Concomitant medication**



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


Concomitant medication is defined as any medication with start date prior to study day 1 and ongoing while on study or any medication with start date on or after study day 1 and up to the end of study.

# Prednisone-equivalent dose

The prednisone-equivalent dose of OCS will be computed based on the table below. Additionally, a multiplier will be applied depending on the dosing frequency: 2 for 'twice daily' or 'every 12 hours' and 0.5 for every other day. For example, cortisone 25 mg is equivalent to prednisone 5 mg and a cortisone 25 mg twice daily is equivalent to prednisone 10 mg/day.

| Corticosteroids | Equivalent dose |
|----------------------------------|-----------------|
| Prednisone | 5 mg |
| Betamethasone | 0.75 mg |
| Cortisone | 25 mg |
| Deflazacort | 6 mg |
| Dexamethasone | 0.75 mg |
| Hydrocortisone | 20 mg |
| Methylprednisolone/Meprednisone/ | 4 mg |
| Methylprednisolone Acetate | |
| Prednisolone | 5 mg |
| Triamcinolone | 4 mg |

# 5.2 Study Points of Reference

#### Baseline

Baseline is the last measurement for the endpoint of interest taken before the first dose of IP. If the measurement is taken on the same day as the first dose and the exact measurement time relative to the first dose is unknown, it will be assumed to have been taken prior to the first dose of IP. If a subject did not receive IP, baseline is the closest recorded measurement on or prior to the randomization date.

#### Study Day 1

Study day 1 for each subject is the first day of IP administration or the day of randomization for subjects who did not receive IP.

# Study Day



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


Study day for each subject is defined as (day of interest – study day 1) + 1 for dates on or after study day 1, or (day of interest – study day 1) for dates prior to study day 1.

#### 5.3 Study Dates

#### **End of 52-Week Treatment Period Date**

End of 52-week treatment period date for each subject is defined as the date of the last assessment for the week 52 visit, the end of study date in case of **subject** early termination, study day 394 **or** (date of study early termination), whichever occurs first.

# **End of Study Date**

End of study for each subject is the date recorded on the End of Study CRF page.

### 5.4 Study Time Intervals

#### **Treatment Period**

The time period from study day 1 to the end of treatment period date inclusive.

# **Final Analysis Period**

The time period from study day 1 to the end of study date, inclusive.

#### 5.5 Arithmetic Calculations

#### Change from baseline

The arithmetic difference between a post-baseline value and baseline for a given timepoint:

(post-baseline value – baseline value).

#### Percent change from baseline

The change from baseline divided by baseline value and multiplied by 100:

(change from baseline / baseline) \* 100.

If the change from baseline is not equal to zero and the baseline value is zero then percent change from baseline is not defined. If the change from baseline is equal to zero and the baseline value is also zero then percent change from baseline is 100.

#### Fold change from baseline or ratio from baseline

Fold change from Baseline equals the post-baseline value divided by the baseline value. If the change from baseline is not equal to 0 and the baseline value is 0 then fold change



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

is not defined. If the change from baseline is equal to 0 and the baseline value is also 0 then fold change is 1.

# 5.6 Efficacy Assessments

# Hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI)

The hSLEDAI is a global index that evaluates disease activity and includes both laboratory and clinical parameters and consists of 24 items. The maximum score is 105. Hybrid SLEDAI is the index score used during the validation of the SLE Responder Index (SRI) (Navarra et al, 2011; Furie et al, 2011). The hSLEDAI includes scleritis and episcleritis in visual disturbance assessments. Scleritis and episcleritis should be confirmed by ophthalmologist and clinically stable if used for scoring purposes. Additionally, arthritis should be scored when > 2 joints manifest signs of inflammation strictly defined as the presence of tenderness plus one of the following: swelling, effusion, warmth or erythema. The presence of tenderness alone is not sufficient and at least 3 joints, and not only 2, must be affected. In this study, for arthritis to be scored it is required to involve the small joints of hands and/or wrists.

Findings should reflect activity during the 30 calendar days prior to the current visit.

Details of hSLEDAI descriptors and the scoring algorithm are described in Appendix B.

#### **British-Isles Lupus Assessment Group (BILAG)**

The BILAG index (BILAG 2004) evaluates disease activity in 9 separate organ systems and comprises a total of 97 items. Each item is measured qualitatively by review of medical history and physical examination (yes/no, improving/same/worse/new) or quantitatively by measuring laboratory values. Based on these items, each of the 9 organ systems allocated an alphabetical score of A (most active), B (moderate activity), C (minor activity), D (stable) or E (never present). The BILAG index can be converted into a numerical score (A grade = 12 points, B = 8, C = 1, D = 0, E = 0). Findings should reflect activity during the 4-week period prior to the current visit and should be related to the subject's SLE. Details of BILAG descriptors and the scoring algorithm are described in Appendix B.

### Physician Global Assessment (PGA) – Visual Analog Scale

The PGA is a visual analog scale (VAS) using 4 descriptive anchors for assessing disease activity over the last 4 weeks. When scoring the PGA VAS, the previous visit score should be noted, and the current score should be relative to that previous visit. The score ranges from 0 to 3 with 3 indicating severe disease. This refers to the most



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

severe possible disease and does not reflect the most severe ever seen in a particular subject, but the most severe disease ever seen in all SLE patients.

This is a global assessment, factoring in all aspects of the subject's lupus disease activity. It should not reflect non-lupus medical conditions. An increase of ≥ 0.3 points (> 10% on the 3 point-VAS) from baseline is considered clinically significant worsening of disease.

# Systemic Lupus Erythematosus Responder Index (SRI-4)

A subject achieves SRI-4 response if all of the following criteria are met:

- 1. ≥ 4-point reduction from baseline in hSLEDAI score
- no new BILAG 2004 A and no > 1 new BILAG 2004 B domain scores compared with baseline (e.g. no B, C, D or E scores at baseline becomes an A or no more than 1 C, D or E score at baseline becomes a B)
- 3. < 0.3-point deterioration from baseline in PGA VAS (scale 0 to 3).
- 4. no use of more than protocol-permitted therapies (i.e. requiring a dose of systemic steroid [for e.g., OCS or intravenous [IV] or intramuscular [IM] corticosteroid] above their baseline dose after week 16; requiring either dose increases of the current immunosuppressants/immunomodulators or initiation of new immunosuppressant/immunomodulatory(s)).

The latest visit date among hSLEDAI, BILAG and PGA VAS will be considered the SRI-4 visit date. In the case when all three visit dates are missing, the upper limit of the analytic window of this visit will be the SRI-4 visit date.

# **BILAG-based Composite Lupus Assessment (BICLA)**

A subject achieves BICLA response if all of the following criteria are met:

- at least one gradation of improvement in baseline BILAG domain scores in all body systems with moderate or severe disease activity at entry (e.g., all A (severe disease) domain scores at baseline falling to B (moderate), C (mild), or D (no activity), and all B domain scores at baseline falling to C or D)
- no new BILAG 2004 A domain score and no > 1 new BILAG 2004 B domain scores compared with baseline
- 3. no worsening of the hSLEDAI score from baseline
- 4. < 0.3-point deterioration from baseline in PGA VAS (scale 0 to 3)



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

5. no use of more than protocol-permitted therapies (i.e. requiring a dose of systemic steroid [for e.g., OCS or IV or IM corticosteroid] above their baseline dose after week 16; requiring either dose increases of the current immunosuppressants/immunomodulators or initiation of new immunosuppressant/immunomodulatory(s)).

# PGA – 4-Point Verbal Rating Scale

The PGA 4-Point Verbal Rating Scale uses 4 verbal descriptors for assessing the severity of disease since the last visit. The options for disease severity are none, mild, moderate, and severe.

This is a global assessment, factoring in all aspects of the subject's lupus disease activity. It should not reflect non-lupus medical conditions. This assessment will be completed by a health care provider (HCP) and must be done before assessing the hSLEDAI and BILAG.

#### Swollen and Tender Joint Count

Joints that have been replaced during the study, or have trauma or received intraarticular injections are considered non-evaluable throughout the study.

Swollen Joint Count Assessments – A total 28 joints will be scored for presence or absence of swelling. A separated score for joints in the hands and wrists will be calculated.

Tender Joint Count Assessments – A total 28 joints will be scored for presence or absence of tenderness. A separated score for joints in the hands and wrists will be calculated.

Swollen and Tender Joint Count Assessments: joints in hands and wrists will be scored for the simultaneous presence or absence of swelling and tenderness.

# Cutaneous Lupus Erythematosus Area and Severity Index (CLASI)

The CLASI consists of 2 scores, the first summarizes the activity of the disease while the second is a measure of the damage done by the disease. Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. Damage is scored in terms of dyspigmentation and scarring, including scarring alopecia. Subjects are asked whether dyspigmentation due to cutaneous lupus lesion usually remains visible for more than 12 months, which is taken to be permanent. If so, the dyspigmentation score is doubled. The scores are calculated



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


by simple addition based on the extent of the symptoms. The CLASI is designed as a table where the rows denote anatomical areas, while the columns score major clinical symptoms. The extent of involvement for each of the skin symptoms is documented according to specific anatomic areas that are scored according to the worst affected lesion within that area for each symptom.

A CLASI response is defined as ≥ 50% improvement of CLASI activity score from baseline.

# **Lupus Low Disease Activity State (LLDAS)**

A subject achieves LLDAS response if all of the following criteria are met:

- hSLEDAI ≤ 4 with no activity in major organ systems (renal [proteinuria, haematuria, pyuria, urinary casts], central nervous system (CNS) [seizure, psychosis, organic brain syndrome, cranial nerve disorder, CVA], cardiopulmonary [pericarditis, pleurisy], vasculitis, fever)
- 2. no new lupus disease activity (i.e. no new descriptor scores in hSLEDAI) compared with the previous assessment
- 3. PGA VAS (scale 0-3) ≤1
- 4. Current prednisolone (or equivalent) dose ≤ 7.5 mg/day
- 5. Standard maintenance doses of immunosuppressive drugs and approved biological agents (i.e. no increase or initiation of immunosuppressive drugs).

#### **BILAG Flare Index**

The BILAG flare index will be derived from BILAG 2004, as measured by BILAG score designation of "worse" or "new" resulting in a B score in ≥ 2 organs or an A score in ≥ 1 organ at one visit (Gordon et al, 2003) compared with the previous available assessment.





Product: Efavaleukin Alfa Protocol Number: 20200234 Date: 25 September 2023






Product: Efavaleukin Alfa
Protocol Number: 20200234

Protocol Number: 20200234

Date: 25 September 2023 

#### Anti-dsDNA

Anti-dsDNA is categorized as negative, indeterminate or positive as follows:

Positive: > 15 IU/mL for subjects in Asia (Japan, Hong Kong, Taiwan and South Korea) and > 75 IU/mL for all other subjects.

Indeterminate: 10 - 15 IU/mL for subjects in Asia (Japan, Hong Kong, Taiwan and South Korea) and 30 - 75 IU/mL for all other subjects.

Negative: < 10 IU/mL for subjects in Asia and < 30 IU/mL for all other subjects.

# 5.7 Patient-reported Outcome (PRO) Assessments Medical Outcomes Short Form-36 Questionnaire Version 2 (SF36v2)

The SF-36v2 (acute version) Health Survey (Ware et al, 2000) contains 36 items and is a revised version of the SF-36 Health Survey. The SF-36v2 acute version is a patient reported generic measure of health status. This survey yields assessments of 8 domains of health-related quality of life: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. The scores from the 8 domains will be evaluated independently and aggregated into 2 norm-based summary component measures of physical and mental health. The recall period is the past 7 days. The scoring of SF-36v2 will be processed by QualityMetric's PRO CoRE Software.

# Patient-Reported Outcome Measurement Information System Fatigue Short Form 7a Instrument (PROMIS Fatigue SF 7A v1.0)

The PROMIS Fatigue Short Form 7a is a 7-item instrument originally constructed by the PROMIS Fatigue team to represent the range of the fatigue trait (PROMIS Fatigue Scoring Manual). It assesses the experience of fatigue as well as its impact on physical, mental and social activities. Both psychometric properties and clinical input were used in the development of the short form from the PROMIS item bank. Estimates of responsiveness and minimally important differences have been reported for the 4 item PROMIS Fatigue instrument in SLE patients (Katz et al, 2019). The PROMIS Fatigue



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023 

has also been able to differentiate disease activity in other rheumatologic diseases. (Wohlfahrt et al, 2019),

Details of the scoring algorithm are described in Appendix C.

# LupusQoL Score

The LupusQoL is the US version of the 34-item PRO originally developed in the United Kingdom (McElhone et al, 2007) for use in adults. This is a SLE-specific health-related quality of life instrument. The LupusQoL consists of 8 domains: physical health (8 items), pain (3 items), planning (3 items), intimate relationships (2 items), burden to others (3 items), emotional health (6 items), body image (5 items), and fatigue (4 items). The final instrument has demonstrated good internal reliability (Cronbach's 0.88 to 0.95), good test-retest reliability (r 0.72 to 0.93), good concurrent validity with the comparable domains of the SF-36 (r 0.71 to 0.79) and good discriminant validity for different levels of disease activity, measured by BILAG index, and damage (Systemic Lupus International Collaborating Clinics/ACR damage index) but not for all domains. The instrument also has acceptable ceiling effects and minimal floor effects.

Details of the scoring algorithm are described in Appendix C.

# **Symptom Questionnaire**

The Symptom Questionnaire is a new patient reported outcome instrument to evaluate inflammatory symptoms, non-inflammatory symptoms, and flare (Pisetsky et al, 2019). The items are based on a 11-point numerical rating scale, with 1 item being a choice of yes or no, all with a 7-day recall. Response to therapy and psychometric properties of the questionnaire will be evaluated with data derived from this study.





Protocol Number: 20200234

Date: 25 September 2023




# 6. Analysis Sets

Product: Efavaleukin Alfa

# 6.1 Full Analysis Set

The Full Analysis Set (FAS) includes all randomized subjects. Data will be analyzed based on randomized treatment assignment.

# 6.2 Safety Analysis Set

The Safety Analysis set includes all randomized subjects who received at least 1 dose of investigational product. Data will be analyzed according to actual treatment received.

# 6.3 Interim Analyses Set(s)

The Interim Analyses Sets include all subjects randomized on or before the interim analyses cutoff dates, and had the opportunity to complete week 16 (actual week 16 visit date ≤ the cutoff date, or randomization date + 126 -1 < the cutoff date). The interim data cutoff dates are based on the number of subjects having the opportunity to complete week 24 visit presented in Table 3-1.



# 7. Planned Analyses

# 7.1 Interim Analysis and Early Stopping Guidelines

Interim analyses will be conducted to inform adaption of the randomization ratio to enroll future subjects to the 3 efavaleukin alfa treatment groups, holding the allocation to placebo constant at 25%, and to assess efficacy for early futility or administrative success decisions:



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


 Data will be subject to ongoing checks for integrity, completeness and accuracy in accordance with the Data Management Plan with the expectation that outstanding data issues are resolved ahead of the snapshot to the extent possible. All available data up to and including the data cut-off date will be included in the analysis based on an "as-is" snapshot of the database without data locking.

- The study team, investigators, and subjects will remain blinded to the results of the IAs unless futility is determined.
- The first IA will be executed after the first 40 subjects are randomized and have had the opportunity to complete the week 24 assessment. Subsequent IAs are scheduled after every additional 32 subjects are randomized and have had the opportunity to complete the week 24 assessment until full enrollment. The last IA will occur when all 320 subjects are randomized and have had the opportunity to complete the week 24 assessment. This IA will be referred to as the 'all-subjects-week-24 IA'.
- Efficacy analyses will be performed at the IAs to assess the likelihood of each
  efavaleukin alfa treatment group being superior to placebo by a clinically meaningful
  difference.
  - From the second IA until before the last IA, if this likelihood is unacceptably low for all dose levels, the trial is recommended to stop for futility.
  - At the 'all-subjects-week-24 IA', if this likelihood is sufficiently high with at least 1 efavaleukin alfa dose level, the IA triggers an administrative success signal. This would not alter ongoing or planned activities of this phase 2b study, but downstream planning for subsequent trials (e.g., a phase 3 study) may commence. Analysis planned each IA are listed in Table 3-1. This interim analysis was cancelled due to the study being terminated for futility prior to the enrollment trigger for this analysis.

#### At IAs:

• For all IAs before full enrollment, the randomization ratio to each active treatment group is proportional to the posterior probability that each group has the highest response rate among the three active treatment groups with power scale of 2.

$$Allocation_d \propto \Pr\left(p_{d,52} = \max_c p_{c,52} \mid \text{Interim Data}\right), \, c,d \in \{low,medium,high}\}$$
 where  $p_{d,52}$  is the posterior probability of achieving SRI-4 response for group d, calculated using a Bayesian independent logistic model with non-informative priors.



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


From the second IA until before the last IA, interim futility analysis will be performed based on the Bayesian Hierarchical Model (BHM) as described in the primary efficacy analysis. Enrollment to the study may be stopped for futility if the posterior probability of achieving a clinically meaningful difference in SRI-4 response rates of at least 15% between each active treatment group and placebo is below 2.5% for all 3 efavaleukin alfa doses.

 $\max \Pr \big( \, p_{d,52} - p_{placebo,52} > \delta \mid \text{Interim Data} \, \, \big) < 0.025, d \in \{low, medium, high\} \\ \text{where } \delta = 0.15 \text{ and } p_{d,52} \text{ is the posterior probability of achieving SRI-4 response for group d, calculated using a BHM.}$ 

• The futility rule and the administrative success trigger are made using estimates of the response rate  $p_{d,52}$  for each dose. However, due to the covariate adjustment, the Bayesian models provide estimates of  $p_d \mid Z$ , the response rate in each dose conditional on the stratification factor Z. The population level estimate for each dose is obtained using a weighted average of the response rate in each stratification group.

$$p_d = \sum_{Z \in Z} w_z \cdot p_d \mid Z \quad \text{for } d \in \{placebo, low, medium, high}\}$$

The set Z indicates the four possible stratification combinations (hSLEDAI stratification [ $\geq$ 10, <10] and region [North America + Western Europe + Asia Pacific vs ROW]). The weights  $w_Z$  will be set equal to the observed proportion of patients in each stratification group at the time of the analysis.

To address the challenge of the lag time between randomization and the week 52 outcome in the adaptive design, a longitudinal model is used to impute week 52 outcome for subjects not yet complete week 52 using their week 16, week 20, or week 24 response data.

# 7.2 Final Analysis

The final analysis will occur after all subjects reach the end of study.

Data will be subject to ongoing checks for integrity, completeness and accuracy in accordance with the Data Management Plan with the expectation that outstanding data issues are resolved ahead of the lock. The data supporting the final analysis will be locked to prevent further changes.



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


# 8. Data Screening and Acceptance

# 8.1 General Principles

The objective of the data screening is to assess the quantity, quality, and statistical characteristics of the data relative to the requirements of the planned analyses.

# 8.2 Data Handling and Electronic Transfer of Data

The Amgen Global Study Operations-Data Management (GSO-DM) department will provide all data to be used in the planned analyses. This study will use the RAVE database. All laboratory, PK, and biomarker data from the central laboratory or vendor will be transferred to GSO-DM. SLE efficacy assessment and PRO data from the central vendor will be transferred to GSO-DM. All other data will be captured on the eCRF.

# 8.3 Handling of Missing and Incomplete Data

Subjects may have missing specific data points for a variety of reasons. In general, data may be missing due to a subject's early withdrawal from study, a missed visit, or non-evaluability of a specific clinical or laboratory measurement at its planned clinical visit.

Additionally, as the study was terminated before the planned completion, subjects may have missed clinical visits including not completing the week 52 visit. For efficacy and PRO outcomes, subjects who terminated early due to sponsor decision will be excluded from analyses of data from visits for which they did not have the opportunity to participate in by the date of study termination decision being communicated to sites, i.e. April 5, 2023. Efficacy data collected after this date will be censored and excluded from analyses for that particular visit. Unless specified, no imputation will be used. The general procedures outlined below describe what will be done when a data point is missing.

#### Hybrid SLEDAI

In case of completely missing hSLEDAI assessment (e.g. missed visit) or partially missing (e.g. laboratory measurements not available), the missing post-baseline hSLEDAI total score will be imputed using last observation carried forward (LOCF) if the previous analysis visit is not missing. Baseline hSLEDAI will not be carried forward to post-baseline.

The hSLEDAl total score will then be computed based on the non-missing and imputed data. If the hSLEDAl total score cannot be evaluated after imputation, the hSLEDAl score ≥ 4 points reduction from baseline will be considered not met.



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


#### CLASI

In case of completely missing CLASI assessment (e.g. missed visit) or partially missing, the missing post-baseline CLASI items will be imputed using LOCF if the previous analysis visit is not missing. Baseline CLASI will not be carried forward to post-baseline.

The CLASI activity score will then be computed based on the non-missing and imputed data. If the CLASI activity score cannot be evaluated after imputation, the CLASI activity score ≥ 50% improvement endpoint will be considered not met.

#### **BILAG**

In case of completely missing BILAG assessment (e.g. missed visit), the missing post baseline BILAG item scores will be imputed using LOCF if the previous analysis visit is not missing.

In case of partially missing, missing laboratory items (e.g. UPCR, creatinine, etc.) will be imputed using LOCF if the previous visit is not missing; other missing items (e.g. active nephritis, Coombs' test positive, etc.) will be imputed as 'No' or 'Not Present'.

Baseline BILAG will not be carried forward to missing post-baseline BILAG.

The BILAG organ domain scores will be calculated based on the non-missing and imputed components. If the non-missing and imputed components are not sufficient to identify the organ domain score, worst scenario approach will be used to determine the BILAG organ domain scores.

#### **PGA VAS**

Missing post-baseline PGA score will be imputed using LOCF if the score at the previous analysis visit is not missing. Baseline PGA will not be carried forward to missing post-baseline PGA.

# SRI-4, BICLA and LLDAS

The criteria for SRI-4, BICLA and LLDAS responses will be evaluated based on the non-missing and imputed PGA, hSLEDAI and BILAG data. If any criteria based on the non-missing and imputed PGA, hSLEDAI and BILAG data cannot be evaluated, then the subject will be considered as a non-responder.

#### **BILAG Flare index**



Product: Efavaleukin Alfa Protocol Number: 20200234

Date: 25 September 2023 

BILAG flare index will be evaluated based on BILAG scores. In case of partially missing BILAG assessment, imputed BILAG scores will be used. In case of

completely missing BILAG assessment, BILAG flare index will remain missing.

**Tender and Swollen Joint Counts** 

If a joint is excluded (non-evaluable or missing), the joint counts will be prorated based

on the algorithm described below.

Prorated Joint Counts: If at least half but not all joints are evaluable (at least 14 joints for

the total 28 joint count, at least 11 joints for the 22 hands and wrists joint count) then the

observed prorated tender or swollen joint count will be calculated. The prorated scores

will be adjusted based upon the number of evaluable joints: the counted score will be

multiplied by 28 (for total) or 22 (for hands and wrists) as applicable and divided by the

number of joints evaluated. If less than half of the joints are evaluable, the number of

tender or swollen joints is missing. For example, if only 25 of the 28 joints are assessed

at a visit and 10 of those 25 are tender/painful and 8 of those 25 are swollen, the

prorated total joint counts are:

Tender: (10/25)\*28 = 11.20,

Swollen: (8/25)\*28 = 8.96.

That is, the values of 11.20 and 8.96 will be used in calculating the % reductions in total

joint counts, not the values of 10 and 8. Similar proration will be conducted for hands

and wrists joint count.

If the tender and swollen joint counts cannot be evaluated after proration, the

tender and swollen joint count ≥ 50% improvement from baseline endpoint will be

considered not met.

Lupus anticoagulant

Lupus anticoagulant results will be derived as follows:

When activated partial thromboplastin time (aPTT) ≤ 29.4 seconds, then

lupus anticoagulant is 'negative'.

When aPTT ≥ 29.4 seconds and hexagonal phospholipid < 11 seconds, then</li>

lupus anticoagulant is 'negative'.

When aPTT ≥ 29.4 seconds and hexagonal phospholipid ≥ 11 seconds, then

lupus anticoagulant is 'positive'.



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


Lupus anticoagulant results will only be derived for baseline, week 24 and week 52 visits.

#### **Dates**

Missing and incomplete dates will be imputed as outlined in Appendix E.

# **Laboratory Toxicity Grading**

In cases when supplemental information for laboratory toxicity grading is missing or the result is ambiguous, the worse toxicity grade possible will be assigned.

# **Laboratory Measurements**

Laboratory measurements that are below the lower quantification limits will be considered equal to the lower limit of quantification for all analyses unless explicitly noted otherwise.

#### 8.4 Detection of Bias

Important protocol deviations and early withdrawal from treatment and from study may bias the results of the study. The incidence of these factors will be assessed and reason for early withdrawals will be tabulated.

# 8.5 Outliers

Scatter plots will be examined to identify potential outliers in any of the continuous variables and frequencies of the categorical data will be examined to identify questionable values. The validity of any questionable values will be verified, and observations found to be due to data entry errors will be queried. Potential outliers that are not due to data entry error will be included in the analysis.

#### 8.6 Distributional Characteristics

Not applicable.

# 8.7 Validation of Statistical Analyses

Programs will be developed and maintained, and output will be verified in accordance with current risk-based quality control procedures.

Tables, figures, and listings will be produced with validated standard macro programs where standard macros can produce the specified outputs.

The production environment for statistical analyses consists of Amgen-supported versions of statistical analysis software; for example, the SAS System version 9.4 or later.



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


# 9. Statistical Methods of Analysis

### 9.1 General Considerations

All categorical variables will be summarized using the number and percent of subjects falling into each category and all continuous variable will be summarized using mean, standard error (SE), standard deviation (SD), median, first quartile (Q1), third quartile (Q3), minimum, maximum, and number of subjects with observations. Safety endpoints will be summarized descriptively, including treatment-emergent adverse events and serious adverse events, clinically significant changes in laboratory values and vital signs, and incidence of antidrug antibodies. All safety analyses will be performed using the Safety Analysis Set based on subject's actual treatment received.

# 9.2 Subject Accountability

The study dates for the first subject enrolled, last subject enrolled, last subject's end of IP **and** last subject's end of study will be presented.

The number and percent of subjects who were randomized, received investigational product, completed investigational product, discontinued investigational product and reasons for discontinuing, completed study, discontinued study and reasons for discontinuing study will be summarized overall and by randomized treatment group. Summary of subjects who discontinue investigational product/study due to COVID-19 control measures will be included.

# 9.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined by the study team before the first subject's initial visit and updated during the IPD reviews throughout the study prior to database lock. These definitions of IPD categories, subcategory codes, and descriptions will be used during the course of the study. Eligibility deviations are defined in the protocol. The final IPD list will be used to produce the summary of IPDs table and the list of subjects with IPDs. IPDs related to COVID-19 control measures will be summarized separately.

# 9.4 Demographic and Baseline Characteristics

The following demographic, baseline characteristics, baseline disease characteristics and baseline therapies of interest will be summarized descriptively by randomized treatment group.

Demographics:

sex (female, male)



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


- age (years)
- age groups ( $\geq$  18 to < 50,  $\geq$  50 and 18 64, 65 74,75 84)
- race (American Indian or Alaska Native, Asian, Black or African-American, Native Hawaiian or Other Pacific Islander, White, Other)
- ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- geographic region (North America [Canada and United States] + Western Europe [Austria, France, Switzerland] + Asia Pacific [Hong Kong, Japan, South Korea and Taiwan], ROW [Bulgaria, Chile, Colombia, Greece, Italy, Mexico, Poland, Russia, Spain and Turkey])

#### Baseline characteristics:

- height (cm)
- weight (kg)
- body mass index (BMI) (kg/m²)

# Baseline disease characteristics:

- years since SLE diagnosis
- hSLEDAI score (continuous, < 10 or ≥ 10)</li>
- baseline hSLEDAI organ involvement (CNS [seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident], vascular [vasculitis], renal [urinary casts, hematuria, proteinuria, pyuria], musculoskeletal [arthritis, myositis], serosal [pleurisy, pericarditis], dermal [rash, alopecia, mucosal ulcers], immunologic [low complement, increased DNA binding], constitutional [fever], hematologic [thrombocytopenia, leukopenia])
- baseline BILAG domain score (A, B, C, D, E)
  - constitutional
  - mucocutaneous
  - neuropsychiatric
  - o musculoskeletal
  - cardiorespiratory
  - gastrointestinal



Product: Efavaleukin Alfa Protocol Number: 20200234

Date: 25 September 2023 

- ophthalmic
- renal
- haematological
- CLASI activity score (continuous, 0, > 0 to  $< 8, \ge 8$ )
- total swollen and tender joint counts
- hand and wrist swollen and tender joint counts
- PGA VAS score
- baseline biomarkers
  - antinuclear antibody (≥ 1:80 vs. negative or < 1:40)
  - anti-dsDNA (continuous, positive, indeterminate or negative)
  - C3, C4 complement (continuous, low or normal/high, low C3 or C4 vs. normal/high C3 and C4)
  - anti-dsDNA and complement
    - o anti-dsDNA positive and low complement
    - anti-dsDNA positive and normal/high complement
    - o anti-dsDNA indeterminate and low complement
    - anti-dsDNA indeterminate and normal/high complement
    - anti-dsDNA negative and low complement
    - anti-dsDNA negative and normal/high complement

#### Baseline medications

- immunosuppressant/immunomodulator (yes, no)
  - mycophenolate mofetil
  - o azathioprine
  - methotrexate
  - anti-malarial (hydroxychloroquine, chloroquine, quinacrine)
  - o dapsone
  - o other
- daily OCS dose (prednisone-equivalent mg/day; continuous, 0 mg/day, > 0 to < 10 mg/day, ≥ 10 mg/day)



Product: Efavaleukin Alfa
Protocol Number: 20200234
Date: 25 September 2023


# 9.5 Efficacy Analyses

Unless stated otherwise, the Full Analysis Set (FAS) will be used for analysis of efficacy endpoints. The efficacy analyses are summarized in Table 9-1, Table 9-2 and Table 9-3.

The SLE efficacy assessment data (BILAG, hSLEDAI, PGA, CLASI, swollen and tender joint counts, **and**) will be submitted to an external independent committee comprised of clinicians with expertise in managing and assessing SLE disease and clinical trials for adjudication. The committee will adjudicate the data and determine whether the efficacy assessments are scored correctly and consistently based on the instruments' specifications.

Unless stated otherwise, the analysis of the SLE efficacy assessment data and their derived endpoints (SRI-4, BICLA, LLDAS and BILAG flare index) will be based on the data resulting from the adjudication. Additionally, to assess the concordance between the investigators and adjudicators, the SRI-4 responses at week 16, 20, 24 and 52 based on the two sources will be cross-tabulated and the concordance rate will be computed as the frequency of cases where the data based on the investigator's assessment and the data resulting from adjudication agree on classification of a subject as an SRI-4 responder/non-responder. If the concordance rate at week 52 is < 0.95, the primary endpoint may be summarized using SRI-4 responses derived based on the investigator-reported data as a sensitivity analysis.


**Table 9-1. Primary Efficacy Endpoint Summary Table** 

| Endpoint | Primary Summary and<br>Analysis Method | Sensitivity and<br>Supplementary Analysis |
|---|---|---|
| SRI-4 response at week 52 | Within each treatment arm, the number and percentage of subjects achieving SRI-4 will be computed. | To assess different data sources: The primary analysis may be repeated using SRI-4 responses based on the investigator data, if the concordance rate is <0.95. |

**Table 9-2. Secondary Efficacy Endpoint Summary Table** 

| Endpo | int | Primary Summary and Analysis Method |
|---|---|---|
| • | BICLA response at week 52 LLDAS response at week 52 Reduction of OCS to ≤ 7.5 mg/day by week 44 and sustained through week 52 in subjects with a baseline OCS dose ≥ 10 mg/day SRI-4 response at week 24 BICLA response at week 24 HSLEDAI reduction ≥ 4 points from baseline at week 24 HSLEDAI reduction ≥ 4 points from baseline at week 52 | Number and percentage of subjects achieving response of interest will be summarized by randomized treatment arm. |
| • | Improvement from baseline in tender and swollen joint count ≥ 50% at weeks 8, 12, 24, 36, and 52 in subjects with ≥ 6 tender and swollen joints involving the hands and wrists at baseline CLASI activity score ≥ 50% improvement from baseline at week 12, 24, 36, and 52 in subjects with a CLASI activity score ≥ 8 at baseline | Number and percentage of subjects achieving response of interest will be summarized by randomized treatment arm. |
| • | Annualized flare rate (as measured by BILAG score designation of "worse" or "new" resulting in a B score in ≥ 2 organs or an A score in ≥ 1 organ) over 52 weeks | Descriptive statistics will be summarized by randomized treatment arm. |
| • | Change from baseline in fatigue standardized score using the PROMIS Fatigue SF 7a at week 12, 24, 36, and 52 Change from baseline in the physical component score, mental | Descriptive statistics will be summarized by randomized treatment arm. |



component score and individual domains of the SF 36 v2 at week 12, 24, 36, and 52

 Change from baseline in the domain scores on the Lupus QoL at weeks 12, 24, 36, and 52

**Table 9-3. Exploratory Efficacy Endpoint Summary Table** 



#### 9.6 Safety Analyses

Product: Efavaleukin Alfa

In the safety analysis, data up to the end of study will be summarized in the final analysis.

#### 9.6.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) version **26.0** or later will be used to code all events categorized as adverse events to a system organ class and a preferred term. The severity of each event will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.

The subject incidence of adverse events will be summarized for all treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation of investigational product, fatal adverse events, treatment-related adverse events, treatment-related serious adverse events, treatment-related adverse events leading to withdrawal of IP, treatment-related fatal adverse events, and adverse events of interest. Subject incidence of treatment-emergent adverse events identified by COVID-19 standardized MedDRA queries and serious adverse events occurring on or after the COVID-19 infection will also be summarized.

Subject incidence of all treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation of investigational product, and fatal adverse events will be tabulated by system organ class in alphabetical order and preferred term in descending order of frequency.

Subject incidence of events of interest (standardized MedDRA queries and/or Amgen Medical Queries) will also be summarized according to their categories and preferred term. Events of interest could include but are not limited to hypersensitivity, tachyarrhythmias, tachypnea, hematopoietic cytopenia, eosinophilic disorder, leucocyte changes, infection and infestation, cytokine release syndrome injection site reaction and drug related hepatic disorder. Number of episodes and duration of treatment-emergent injection site reactions will be further summarized by treatment group.

Overall summary of subject incidence of treatment-emergent adverse events and by preferred term and worst severity grade will be provided by anti-AMG592 and Anti-IL-2 antibody status.



Summaries of treatment-emergent and serious adverse events will be tabulated by system organ class, preferred term, and grade. An overall summary of adverse events by **severity** grade will be provided.

Summary of exposure-adjusted subject rates of treatment-emergent adverse events will be tabulated overall and by system organ class and preferred term.

#### 9.6.2 Laboratory Test Results

Selected clinical laboratory test results, presented in Table 9-4, change and percent change from baseline will be summarized over time by each treatment group. In addition, shift tables, from baseline to the worst on-study laboratory toxicity based on the CTCAE version 5, will be presented.

Subject incidence of worst post-baseline of eosinophils counts and percentages by the laboratory normal range will be tabulated by treatment group.

Table 9-4 Selected Safety Laboratory Tests

| Central Laboratory: | Central Laboratory: Urinalysis |
|---|---|
| Hematology | |
| RBC | Protein/creatinine ratio |
| Hemoglobin | |
| Hematocrit | |
| Platelets | |
| Reticulocytes | |
| WBC | |
| Differential | |
| <ul> <li>Eosinophils</li> </ul> | |
| <ul> <li>Lymphocytes</li> </ul> | |
| Total neutrophils | |
| | Hematology RBC Hemoglobin Hematocrit Platelets Reticulocytes WBC Differential • Eosinophils • Lymphocytes |

ALP = alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate aminotransferase; CK = creatinine kinase; GGT = gamma glutamyl transferase; MDRD = Modification of Diet in Renal Disease; RBC = red blood cell count; WBC = white blood cell count

#### 9.6.3 Vital Signs

The actual value, change and percent change from baseline in vital signs will be summarized over time by treatment arm for diastolic blood pressure **and**, heart rate.

#### 9.6.4 Electrocardiogram

The electrocardiogram (ECG) measurements from this clinical study were performed as per standard of care for routine safety monitoring, rather than for purposes of assessment of potential QT interval corrected (QTc) effect. Because these evaluations may not necessarily be performed under the rigorous conditions expected to lead to meaningful evaluation of QTc data; neither summaries nor statistical analyses will be



provided, and these data would not be expected to be useful for meta-analysis with data from other trials.



#### 9.6.6 Exposure to Investigational Product

Descriptive statistics will be produced to describe the exposure to IP by treatment arm. Summary statistics will be provided for the total dose received and total duration of IP exposure by treatment arm.

#### 9.6.7 Exposure to Other Protocol-permitted Therapy

Other protocol-required therapies for this study are immunomodulators/immunosuppressants, OCS, NSAIDs, topical corticosteroids and topical calcineurin inhibitors and anti-proteinuria agents.

The baseline exposure to OCS and immunomodulators/immunosuppressants will be summarized using descriptive statistics (number and percentages).

## 9.6.8 Exposure to Concomitant Medication

Not applicable.

#### 9.7 Other Analyses

Medical history will be summarized by SOC and PT and tabulated by treatment group and total using the Safety Analysis Set according to the actual treatment received.

### 9.7.1 Analyses of Pharmacokinetic Endpoints

Amgen Clinical Pharmacology Modeling and Simulation (CPMS) group will conduct PK analysis. Serum concentration data will be summarized by treatment for each PK sampling time point. PK parameters may be summarized if adequately estimated.

The descriptive statistics for absolute change from baseline, percentage change from baseline and ratio to baseline will be provided by treatment arms at specified time-points for the endpoints C3, C4, anti-dsDNA antibody and antiphospholipid



**Date: 25 September 2023** 

antibody (anticardiolipin antibody IgG and IgM, beta-2 glycoprotein IgG and IgM and lupus anticoagulant).

#### 9.7.2 Analyses of Clinical Outcome Assessments

The PRO endpoints include fatigue standardized score using PROMIS Fatigue SF 7, physical and mental component score and individual domains of the SF 36 v2.

#### 9.7.3 Analyses of Biomarker Endpoints

Exploratory biomarker analyses beyond those mentioned in this SAP may be conducted by Amgen Clinical Biomarker group.

#### 10. Changes From Protocol-specified Analyses

Based on the Data Monitoring Committee's recommendation after interim analysis 3 and subsequent decision by the Data Access Plan Team, enrollment in the study was stopped and the study terminated as the study met the pre-specified futility criteria. As such, some analyses that were initially planned in the protocol will not be performed. Key changes from protocol-specified analyses are as follows:

- Removal of subsequent IAs following study early termination.
- Removal of some exploratory endpoints.
- Removal of statistical comparison of treatment groups at the final analysis;
   descriptive statistics by treatment groups will be generated instead.

#### 11. Literature Citations / References

Agresti A. Categorical Data Analysis, New York: John Wiley & Sons, Inc, 1990.

Buyon JP, Petri MA, Kim MY, et. al. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: A randomized trial. Ann Intern Med. 2005;142:953.

Efavaleukin Alfa Investigator's Brochure. Thousand Oaks, CA. Amgen Inc.

Franklyn K, Lau CS, Navarra SV, et al. Definition and initial validation of a Lupus Low Disease Activity State (LLDAS). *Ann Rheum Dis*. 2016 Sep;75(9):1615-1621.

Furie RA, Petri MA, Wallace DJ, et al. Novel evidence-based systemic lupus erythematosus responder index. Arthritis & Rheum. 2009;61(9):1143-1151.

Gladman D, Ginzler E, Goldsmith C, et al. The development and initial validation of the systemic lupus international collaborating clinics/American College of Rheumatology Damage Index for Systemic Lupus Erythematosus. Arthritis Rheum. 1996; 39(3):363-369.

Golder V, Kandane-Rathnayake R, Huq M, et al. Lupus low disease activity state as a treatment endpoint for systemic lupus erythematosus: a prospective validation study. Lancet Rheum. 2019;1(2):e95-e102.

Gordon C, Sutcliffe N, Skan J, et al. Definition and treatment of lupus flares measured by the BILAG index. *Rheumatology*. 2003;42(11):1372-9.



Jolly M, Pickard AS, Wilke C et al. Lupus-specific health outcome measure for US patients: the LupusQoL-US version. Ann Rheum Dis. 2010;69:29-33.

Katz P, Pedro S, Alemao E, et al. Estimates of responsiveness, minimally import differences and patient acceptable symptom state in five patient-reported outcomes measurement information system short forms in systemic lupus erythematosus. ACR Open. 2019: 1-8. Doi 10.1002/acr2.11100

Kenward MG and Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. Biometrics. 1997; 53: 983-997

Khraishi M, Aslanov R, Dixit S, et al 2014. The validity of patient and physician global disease activity assessments of systemic lupus erythematosus: results from the lupus activity coring tool (LAST) as compared to the Selena Sledai (SS) modification multicentre study. *ACR* 2014.

Liang MH, Socher SA, Larson MG, Schur PH. Reliability and validity of six systems for the clinical assessment of disease activity in systemic lupus erythematosus. *Arthritis Rheum.* 1989;32(9):1107-18.

Longford NT. Random Coefficient Models, New York: Oxford University Press, Inc, 1993

McElhone K, Abbott J, Shelmerdine J et al. Development and validation of a disease specific health-related quality of life measure, the LupusQol, for adults with systemic lupus erythematosus. Arthritis Rheum. 2007;57:972-979.

Navarra SV, Guzmán RM, Gallacher AE, et al. Efficacy and safety of belimumab in patients with active systemic lupus erythematosus: a randomised, placebo-controlled, phase 3 trial. *Lancet*. 2011 Feb 26;377(9767):721-731.

Pisetsky DS, Clowse MEB, Criscione-Schreiber LG, et al. A Novel System to Categorize the Symptoms of Systemic Lupus Erythematosus. *Arth Care Res.* 2019;71(6):735-741.

PROMIS Fatigue Scoring Manual. Accessed at http://www.healthmeasures.net/images/PROMIS/manuals/PROMIS\_Fatigue\_Scoring\_M anual.pdf on 29 Jan 2020

Ware JE. SF-36 Health Survey Update. SPINE. 2000; 25:3130-3139.

Wohlfahrt A, Bingham CO, Marder W, et al. Responsiveness of patient-reported outcomes measurement information system measures in rheumatoid arthritis patients starting or switching a disease-modifying antirheumatic drug. Arth Car Res 2019: (4): 521-529.

Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage 1997; 13: 63-74.



#### 12. Appendices

## Appendix A. Reference Values/Toxicity Grades

Assessment of severity for each adverse event and serious adverse event reported during the study will be based on:

The Common Terminology Criteria for Adverse Events (CTCAE), version 5 which is available at the following location:

http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm



## **Appendix B. SLE Assessment Forms/Instruments**

The hSLEDAI score is computed as sum of the score across the descriptors.

| Weight | Score | Descriptor | Definition |
|---|---|---|---|
| 8 | | Seizure | Recent onset, exclude metabolic, infectious or drug causes |
| 8 | | Psychosis | Altered ability to function in normal activity due to severe disturbance in the perception of reality. Include hallucinations, incoherence, marked loose associations, impoverished thought content, marked illogical thinking, bizarre, disorganized or catatonic behavior. Exclude uremia and drug causes |
| 8 | | Organic brain<br>syndrome | Altered mental function with impaired orientation, memory, or other intellectual function, with rapid onset and fluctuating clinical features, inability to sustain attention to environment, plus at least two of the following: perceptual disturbance, incoherent speech, insomnia or daytime drowsiness, or increased or decreased psychomotor activity. Exclude metabolic, infection, or drug causes |
| 8 | | Visual<br>disturbance | Retinal changes of SLE. Include cystoid bodies, retinal hemorrhages, serous exudate or hemorrhages in the choroid, optic neuritis, scleritis or episcleritis. Exclude hypertension, infection, or drug causes |
| 8 | | Cranial nerve disorder | New onset of sensory or motor neuropathy involving cranial nerves |
| 8 | | Lupus<br>headache | Severe, persistent headache; may be migrainous, but must be non-responsive to narcotic analgesia. |
| 8 | | CVA | New onset of cerebrovascular accident(s). Exclude arterisclerosis |
| 8 | | Vasculitis | Ulceration, gangrene, tender finder nodules, periungual infarction, splinter hemorrhages, or biopsy or angiogram proof of vasculitis |
| 4 | | Arthritis | >2 joints of hands and wrists with signs of inflammation (i.e., tenderness with swelling or effusion) |




| 4 | Myositis | Proximal muscle aching/weakness, associated with elevated creatinine phosphokinase (CK)/aldolase or EMG changes or a biopsy showing myositis |
|---|---|---|
| 4 | Urinary casts | Heme-granular or RBC casts |
| 4 | Hematuria | > 5 RBC/high power field. Exclude stone, infection, or other cause |
| 4 | Proteinuria | More than 0.5 gram/24 hours. |
| 4 | Pyuria | > 5 WBC/high power field. Exclude infection |
| 2 | Rash | Inflammatory type rash. |
| 2 | Alopecia | Abnormal, patchy or diffuse loss of hair |
| 2 | Mucosal ulcers | Oral or nasal ulcerations |
| 2 | Pleurisy | Pleuritic chest pain or pleural rub with effusion or pleural thickening . |
| 2 | Pericarditis | Classic pericardial pain and/or rub effusion with ECG confirmation |
| 2 | Low complement | Decrease in CH50, C3, or C4 < lower limit of nl for testing laboratory |
| 2 | Increased DNA binding | Increased DNA binding above normal range for testing laboratory |
| 1 | Fever | > 38 °C. Exclude infectious cause |
| 1 | Thrombocytope nia | < 100 x 10 <sup>9</sup> platelets / L, exclude drug causes. |
| 1 | Leukopenia | < 3 x 10 <sup>9</sup> WBC/L, exclude drug causes |

**BILAG-2004 Index Form** 



#### **BILAG2004 INDEX**

Only record items due to SLE Disease Activity & assessment

| Scoring: ND Not Done | | | CARDIORESPIRATORY | |
|---|---|---|---|---|
| 1 Improving | | | 44. Myocarditis - mild ( | ) |
| 2 Same | | | 45. Myocarditis/Endocarditis + Cardiac failure ( | ) |
| 3 Worse | | | 46. Arrhythmia | ) |
| 4 New | | | 47. New valvular dysfunction ( | ) |
| Yes/No OR Value (where indicated) indicate if not due to SLE activ | | | 48. Pleurisy/Pericarditis (<br>49. Cardiac tamponade ( | , |
| indicate if not due to SLE active (default is 0 = not present) | ity | | 50. Pleural effusion with dyspnoea ( | ( |
| (default is 0 – not present) | | | 51. Pulmonary haemorrhage/vasculitis ( | 1 |
| CONSTITUTIONAL | | | 52. Interstitial alveolitis/pneumonitis ( | í |
| 1. Pyrexia - documented > 37.5°C | ( | ) | 53. Shrinking lung syndrome ( | í |
| <ol><li>Weight loss - unintentional &gt; 5%</li></ol> | è | j . | 54. Aortitis ( | ) |
| 3. Lymphadenopathy/splenomegaly | ( | ) | 55. Coronary vasculitis ( | ) |
| 4. Anorexia | ( | ) | | |
| | | | GASTROINTESTINAL | |
| MUCOCUTANEOUS | | | 56. Lupus peritonitis ( | ) |
| 5. Skin eruption - severe | 9 | , | 57. Abdominal serositis or ascites | ) |
| 6. Skin eruption - mild<br>7. Angio-oedema - severe | 5 | ) | 58. Lupus enteritis/colitis (<br>59. Malabsorption ( | ? |
| 8. Angio-oedema - mild | > | - ( | 60. Protein losing enteropathy ( | < |
| 9. Mucosal ulceration - severe | 7 | - ( | 61. Intestinal pseudo-obstruction ( | ( |
| 10. Mucosal ulceration - mild | 7 | - 1 | 62. Lupus hepatitis | 5 |
| 11. Panniculitis/Bullous lupus - severe | ì | - í | 63. Acute lupus cholecystitis ( | í . |
| 12. Panniculitis/Bullous lupus - mild | è | j . | 64. Acute lupus pancreatitis ( | j . |
| <ol><li>Major cutaneous vasculitis/thrombosis</li></ol> | ( | ) | | |
| <ol> <li>Digital infarcts or nodular vasculitis</li> </ol> | ( | ) | OPHTHALMIC | |
| 15. Alopecia - severe | ( | ) | 65. Orbital inflammation/myositis/proptosis ( | ) |
| 16. Alopecia - mild | ( | ) | 66. Keratitis - severe | ) |
| 17. Peri-ungual erythema/chilblains | 9 | ) | 67. Keratitis - mild | ) |
| 18. Splinter haemorrhages | ( | ) | 68. Anterior uveitis ( | , |
| NEUDOBENCIII (TDIC | | | 69. Posterior uveitis/retinal vasculitis - severe ( 70. Posterior uveitis/retinal vasculitis - mild ( | ? |
| NEUROPSYCHIATRIC 19. Aseptic meningitis | | | 71. Episcleritis ( | ( |
| 20. Cerebral vasculitis | λ | - 1 | 72. Scleritis - severe ( | ( |
| 21. Demyelinating syndrome | 7 | - 5 | 73. Scleritis - mild | 1 |
| 22. Myelopathy | 7 | ś | 74. Retinal/choroidal vaso-occlusive disease ( | í |
| 23. Acute confusional state | è | í | 75. Isolated cotton-wool spots (cytoid bodies) ( | j . |
| 24. Psychosis | | j . | 76. Optic neuritis | j . |
| 25. Acute inflammatory demyelinating | | ) | 77. Anterior ischaemic optic neuropathy ( | ) |
| polyradiculoneuropathy | | | | |
| <ol><li>Mononeuropathy (single/multiplex)</li></ol> | ( | ) | RENAL | |
| 27. Cranial neuropathy | ( | ) | 78. Systolic blood pressure (mm Hg) value ( | ) 🗆 |
| 28. Plexopathy | 9 | ) | 79. Diastolic blood pressure (mm Hg) value ( | ) 🗆 |
| 29. Polyneuropathy<br>30. Seizure disorder | 5 | - { | 80. Accelerated hypertension Yes/No (<br>81. Urine dipstick protein (+=1, ++=2, +++=3) ( | 30 |
| 31. Status epilepticus | } | - ( | 82. Urine albumin-creatinine ratio mg/mmol ( | ( ii |
| 32. Cerebrovascular disease (not due to vasculitis) | 7 | 1 | 83. Urine protein-creatinine ratio mg/mmol ( | ( i |
| 33. Cognitive dysfunction | ì | - í | 84. 24 hour urine protein (g) value ( | ( iii |
| 34. Movement disorder | ( ) | 5 | 85. Nephrotic syndrome Yes/No ( | ) |
| 35. Autonomic disorder | ( | ) | 86. Creatinine (plasma/serum) µmol/1 ( | ) 🗆 |
| 36. Cerebellar ataxia (isolated) | ( | ) | 87. GFR (calculated) ml/min/1.73 m <sup>2</sup> ( | ) 🗆 |
| <ol> <li>Lupus headache - severe unremitting</li> </ol> | ( | ) | 88. Active urinary sediment Yes/No ( | ) |
| 38. Headache from IC hypertension ( ) 89. Active | | 89. Active nephritis Yes/No ( | ) | |
| ARROSET COMPANY | | | H. FM. FOI OCIC. I | |
| MUSCULOSKELETAL<br>39. Myositis - severe | | | HAEMATOLOGICAL<br>90. Haemoglobin (g/dl) value ( | ) 🗆 |
| 40. Myositis - mild | | - ( | 90. Haemoglobin (g/dl) value (<br>91. Total white cell count (x 10 <sup>6</sup> /l) value ( | ) |
| 41. Arthritis ( severe) | | - 5 | 92. Neutrophils (x 10 <sup>9</sup> /l) value ( | 15 |
| 42. Arthritis (moderate)/Tendonitis/Tenosynovitis | | í | 93. Lymphocytes (x 10 <sup>6</sup> /l) value ( | ( ii |
| 43. Arthritis (mild)/Arthralgia/Myalgia | | j . | 94. Platelets (x 10 <sup>6</sup> /l) value ( | ή <u> </u> |
| | | - | 95. TTP | ) |
| Weight (kg): | | 96. Evidence of active haemolysis Yes/No ( | ) | |
| 97. Coombs' test positive (isolated) Yes/N | | 97. Coombs' test positive (isolated) Yes/No ( | ) | |
| Revision: 12/Jan/2007 | | | | |
| | | | 5 · · · · · | |
| Investigator initials: | | | Date of assessment: | |

#### **BILAG-2004 INDEX SCORING**

• scoring based on the principle of physician's intention to treat

| Category | Definition |
|---|---|
| A | Severe disease activity requiring any of the following treatment: 1. systemic high dose oral glucocorticoids (equivalent to prednisolone > 20 mg/day) |



| | <ul> <li>2. intravenous pulse glucocorticoids (equivalent to pulse methylprednisolone ≥ 500 mg)</li> <li>3. systemic immunomodulators (include biologicals, immunoglobulins and plasmapheresis)</li> </ul> |
|---|---|
| | 4. therapeutic high dose anticoagulation in the presence of high dose steroids or immunomodulators |
| В | e.g.: warfarin with target INR 3 - 4 Moderate disease activity requiring any of the following treatment: 1. systemic low dose oral glucocorticoids (equivalent to prednisolone ≤ 20 mg/day) 2. intramuscular or intra-articular or soft tissue glucocorticoids injection (equivalent to methylprednisolone < 500mg) 3. topical glucocorticoids 4. topical immunomodulators 5. antimalarials or thalidomide or prasterone or acitretin 6. symptomatic therapy e.g.: NSAIDs for inflammatory arthritis |
| С | Mild disease |
| D | Inactive disease but previously affected |
| E | System never involved |

## **BILAG Constitutional Scoring Algorithm**

| Grade | Criteria |
|---|---|
| А | <ol> <li>Pyrexia recorded as 2 (same), 3 (worse) or 4 (new) AND</li> <li>Any 2 or more of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>Weight loss</li> <li>Lymphadenopathy/splenomegaly</li> <li>Anorexia</li> </ul> </li> </ol> |
| В | <ol> <li>Pyrexia recorded as 2 (same), 3 (worse) or 4 (new) OR</li> <li>Any 2 or more of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>Weight loss</li> <li>Lymphadenopathy/splenomegaly</li> <li>Anorexia</li> </ul> </li> <li>BUT do not fulfil criteria for Category A</li> </ol> |
| С | <ol> <li>Pyrexia recorded as 1 (improving) OR</li> <li>One or more of the following recorded as &gt; 0: <ul> <li>Weight loss</li> <li>Lymphadenopathy/Splenomegaly</li> <li>Anorexia</li> </ul> </li> </ol> |



| | BUT does not fulfil criteria for category A or B |
|---|---|
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits |
| | or domain previous involvement is yes) |
| E | No previous involvement |
| Missing | |

## **BILAG Mucocutaneous Scoring Algorithm**

| Grade | Criteria |
|---|---|
| А | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): a) Skin eruption - severe b) Angio-oedema - severe c) Mucosal ulceration - severe d) Panniculitis/Bullous lupus - severe e) Major cutaneous vasculitis/thrombosis |
| В | <ol> <li>Any Category A features recorded as 1 (improving) OR</li> <li>Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ol> <li>Skin eruption - mild</li> <li>Panniculitis/Bullous lupus - mild</li> <li>Digital infarcts or nodular vasculitis</li> <li>Alopecia - severe</li> </ol> </li> </ol> |
| С | <ul> <li>a) Any Category B features recorded as 1 (improving) OR</li> <li>b) Any of the following recorded as &gt; 0: <ul> <li>a) Angio-oedema - mild</li> <li>b) Mucosal ulceration - mild</li> <li>c) Alopecia - mild</li> <li>d) Periungual erythema/chilblains</li> <li>e) Splinter haemorrhages</li> </ul> </li> </ul> |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Neuropsychiatric Scoring Algorithm**

| Grade | Criteria |
|---|---|
| A | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): 1. Aseptic meningitis 2. Cerebral vasculitis 3. Demyelinating syndrome 4. Myelopathy 5. Acute confusional state 6. Psychosis 7. Acute inflammatory demyelinating polyradiculoneuropathy 8. Mononeuropathy (single/multiplex) 9. Cranial neuropathy 10. Plexopathy |



| | 11. Polyneuropathy<br>12. Status epilepticus<br>13. Cerebellar ataxia |
|---|---|
| В | <ul> <li>a) Any Category A features recorded as 1 (improving) OR</li> <li>b) Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>a) Seizure disorder</li> <li>b) Cerebrovascular disease (not due to vasculitis)</li> <li>c) Cognitive dysfunction</li> <li>d) Movement disorder</li> <li>e) Autonomic disorder</li> <li>f) Lupus headache - severe unremitting</li> <li>g) Headache due to raised intracranial hypertension</li> </ul> </li> </ul> |
| С | Any Category B features recorded as 1 (improving) |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Musculoskeletal Scoring Algorithm**

| Grade | Criteria |
|---|---|
| А | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): a) Severe Myositis b) Severe Arthritis |
| В | <ol> <li>Any Category A features recorded as 1 (improving) OR</li> <li>Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>Mild Myositis</li> <li>Moderate Arthritis/Tendonitis/Tenosynovitis</li> </ul> </li> </ol> |
| С | Any Category B features recorded as 1 (improving) OR Any of the following recorded as > 0: a) Mild Arthritis/Arthralgia/Myalgia |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Cardiorespiratory Scoring Algorithm**

| Grade | Criteria |
|---|---|
| A | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): a) Myocarditis/Endocarditis + Cardiac failure b) Arrhythmia c) New valvular dysfunction |



| | d) Cardiac tamponade e) Pleural effusion with dyspnoea f) Pulmonary haemorrhage/vasculitis g) Interstitial alveolitis/pneumonitis h) Shrinking lung syndrome i) Aortitis j) Coronary vasculitis |
|---|---|
| В | <ol> <li>Any Category A features recorded as 1 (improving) OR</li> <li>Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>a) Pleurisy/Pericarditis</li> <li>b) Myocarditis - mild</li> </ul> </li> </ol> |
| С | Any Category B features recorded as 1 (improving) |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Gastrointestinal Scoring Algorithm**

| Grade | Criteria |
|---|---|
| A | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): a) Peritonitis b) Lupus enteritis/colitis c) Intestinal pseudo-obstruction d) Acute lupus cholecystitis e) Acute lupus pancreatitis |
| В | <ol> <li>Any Category A feature recorded as 1 (improving) OR</li> <li>Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>a) Abdominal serositis and/or ascites</li> <li>b) Malabsorption</li> <li>c) Protein losing enteropathy</li> <li>d) Lupus hepatitis</li> </ul> </li> </ol> |
| С | Any Category B features recorded as 1 (improving) |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Ophthalmic Scoring Algorithm**



| Grade | Criteria |
|---|---|
| A | Any of the following recorded as 2 (same), 3 (worse) or 4 (new): a) Orbital inflammation/myositis/proptosis b) Keratitis - severe c) Posterior uveitis/retinal vasculitis - severe d) Scleritis - severe e) Retinal/choroidal vaso-occlusive disease f) Optic neuritis g) Anterior ischaemic optic neuropathy |
| В | <ol> <li>Any Category A features recorded as 1 (improving) OR</li> <li>Any of the following recorded as 2 (same), 3 (worse) or 4 (new): <ul> <li>a) Keratitis - mild</li> <li>b) Anterior uveitis</li> <li>c) Posterior uveitis/retinal vasculitis - mild</li> <li>d) Scleritis - mild</li> </ul> </li> </ol> |
| С | <ol> <li>Any Category B features recorded as 1 (improving) OR</li> <li>Any of the following recorded as &gt; 0: <ul> <li>a) Episcleritis</li> <li>b) Isolated cotton-wool spots (cystoid bodies)</li> </ul> </li> </ol> |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

## **BILAG Renal Scoring Algorithm**

| Grade | Criteria |
|---|---|
| A | <ul> <li>Two or more of the following providing 1, 4 or 5 is included:</li> <li>1. Deteriorating proteinuria (severe) defined as <ul> <li>a) urine dipstick increased by ≥ 2 levels (used only if other methods of urine protein estimation not available); or</li> <li>b) 24-hour urine protein &gt; 1 g that has not decreased (improved) by ≥ 25%; or</li> <li>c) urine protein-creatinine ratio &gt; 100 mg/mmol that has not decreased (improved) by ≥ 25%; or</li> <li>d) urine albumin-creatinine ratio &gt; 100 mg/mmol that has not decreased (improved) by ≥ 25%</li> </ul> </li> <li>2. Accelerated hypertension</li> <li>3. Deteriorating renal function (severe) defined as <ul> <li>a) plasma creatinine &gt; 130 μmol/l and having risen to &gt; 130% of previous value; or</li> <li>b) GFR &lt; 80 ml/min per 1.73 m² and having fallen to &lt; 67% of previous value; or</li> <li>c) GFR &lt; 50 ml/min per 1.73 m², and last time was &gt; 50 ml/min per 1.73 m² or was not measured.</li> </ul> </li> </ul> |




| | 4. Active urinary sediment |
|---|---|
| | 5. Histological evidence of active nephritis within last 3 months |
| | 6. Nephrotic syndrome |
| В | <ol> <li>One of the following:</li> <li>One of the Category A feature</li> <li>Proteinuria (that has not fulfilled Category A criteria) <ul> <li>a) urine dipstick which has risen by 1 level to at least 2+ (used only if other methods of urine protein estimation not available); or</li> <li>b) 24-hour urine protein ≥ 0.5 g that has not decreased (improved) by ≥ 25%; or</li> <li>c) urine protein-creatinine ratio ≥ 50 mg/mmol that has not decreased (improved) by ≥ 25%; or</li> <li>d) urine albumin-creatinine ratio ≥ 50 mg/mmol that has not decreased (improved) by ≥ 25%</li> </ul> </li> <li>Plasma creatinine &gt; 130 μmol/l and having risen to ≥ 115% but ≤ 130%</li> </ol> |
| | of previous value |
| С | <ul> <li>One of the following:</li> <li>1. Mild/Stable proteinuria defined as <ul> <li>a) urine dipstick ≥ 1+ but has not fulfilled criteria for Category A &amp; B (used only if other methods of urine protein estimation not available); or</li> <li>b) 24 hour urine protein &gt; 0.25 g but has not fulfilled criteria for Category A &amp; B; or</li> <li>c) urine protein-creatinine ratio &gt; 25 mg/mmol but has not fulfilled criteria for Category A &amp; B; or</li> <li>d) urine albumin-creatinine ratio &gt; 25 mg/mmol but has not fulfilled criteria for Category A &amp; B</li> </ul> </li> <li>2. Rising blood pressure (providing the recorded values are &gt; 140/90 mm Hg) which has not fulfilled criteria for Category A &amp; B, defined as <ul> <li>a) systolic rise of ≥ 30 mm Hg; and</li> <li>b) diastolic rise of ≥ 15mm Hg</li> </ul> </li> </ul> |
| D | Previous involvement (i.e. A, B, C or D domain grade at any previous visits or domain previous involvement is yes) |
| Е | No previous involvement |
| Missing | |

Since the urine albumin-creatinine ratio and 24-hour urine protein are not collected in this study, the criteria for BILAG proteinuria will be based on urine dipstick and urine protein-creatinine ratio only.

## **BILAG Hematological Scoring Algorithm**

| Grade | Criteria |
|---|---|
| A | <ol> <li>TTP recorded as 2 (same), 3 (worse) or 4 (new) or</li> <li>Any of the following: <ul> <li>a) Evidence of haemolysis and Haemoglobin &lt; 8 g/dl</li> </ul> </li> </ol> |



| | b) Platelet count < 25 x 10 <sup>9</sup> /l |
|---|---|
| | 1. TTP recorded as 1 (improving) or |
| | 2. Any of the following: |
| 1_ | a) Evidence of haemolysis and Haemoglobin 8 - 9.9 g/dl |
| В | b) Haemoglobin < 8 g/dl (without haemolysis) |
| | c) White cell count < 1.0 x 10 <sup>9</sup> /l |
| | d) Neutrophil count < 0.5 x 10 <sup>9</sup> /l |
| | e) Platelet count 25 - 49 x 10 <sup>9</sup> /l |
| Any of the following: | |
| | a) Evidence of haemolysis and Haemoglobin ≥ 10g/dl |
| | b) Haemoglobin 8 - 10.9 g/dl (without haemolysis) |
| | c) White cell count 1 - 3.9 x 10 <sup>9</sup> /l |
| С | d) Neutrophil count 0.5 - 1.9 x 10 <sup>9</sup> /l |
| | e) Lymphocyte count < 1.0 x 10 <sup>9</sup> /L |
| | f) Platelet count 50 - 149 x 10 <sup>9</sup> /l |
| | 1) 1 latelet count 30 - 143 x 10 /1 |
| | g) Isolated Coombs' test positive |
| _ | Previous involvement (i.e. A, B, C or D domain grade at any previous visits |
| D | or domain previous involvement is yes) |
| _ | - |
| E | No previous Involvement. |
| Missing | |
| wiiosirig | |

## **LLDAS**

| Criteria | Derivation |
|---|---|
| HSLEDAI ≤ 4 with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) | HSLEDAI score ≤ 4 proteinuria, haematuria, pyuria, urinary casts, seizure, psychosis, organic brain syndrome, cranial nerve disorder, CVA, pericarditis, pleurisy, vasculitis and fever in hSLEDAI are marked 'not present' |
| No new lupus activity compared with the previous assessment | No new 'present' hSLEDAI descriptors compared to previous visit |
| PGA ≤ 1 | PGA ≤ 1 |



| Current prednisolone (or equivalent) dose ≤ 7.5 mg/day | Prednisone equivalent is ≤ 7.5 mg/day at the visit |
|---|---|
| Standard maintenance doses of immunosuppressive drugs and approved biological agents (i.e. no increase or initiation of immunosuppressive drugs.) | No new or increase in immunosuppressant at the visit |

## Appendix C. Patient-reported Outcome Forms/Instruments

#### C1. SF-36 Version 2

SF-36 items will be scored using the SF-36 version 2.0 Quality Metric Health Outcome Scoring Software (Ware et al, 2007).

#### C2. Scoring algorithm for PROMIS Fatigue SF 7A

PROMIS SF v1.0 – Fatigue 7A will be scored according to the PROMIS Fatigue Brief Guide including the scoring in the Instrument Section downloaded from

http://www.healthmeasures.net/images/PROMIS/manuals/PROMIS Fatigue Scoring M anual.pdf on 28 Feb 2019.

To calculate the score for PROMIS Fatigue SF 7A, sum the values of the responses to each of the 7 questions. The lowest and highest possible sum is 7 and 35, respectively. Then, use the table below to rescale the score into a standardize score with a mean of 50 and a standard deviation of 10.

| Conversion Table | |
|------------------|---------|
| Raw score | T-score |
| 7 | 29.4 |
| 8 | 33.4 |
| 9 | 36.9 |
| 10 | 39.6 |
| 11 | 41.9 |
| 12 | 43.9 |
| 13 | 45.8 |
| 14 | 47.6 |
| 15 | 49.2 |
| 16 | 50.8 |
| 17 | 52.2 |
| 18 | 53.7 |
| 19 | 55.1 |
| 20 | 56.4 |
| 21 | 57.8 |
| 22 | 59.2 |
| 23 | 60.6 |
| 24 | 62.0 |
| 25 | 63.4 |



| 26 | 64.8 |
|----|------|
| 27 | 66.3 |
| 28 | 67.8 |
| 29 | 69.4 |
| 30 | 71.1 |
| 31 | 72.9 |
| 32 | 74.8 |
| 33 | 77.1 |
| 34 | 79.8 |
| 35 | 83.2 |

#### C3. Scoring algorithm for Modified LupusQoL

The LupusQoL will be scored using the scoring algorithm from the RWS Life Science website accessed 10 April 2020. http://www.corptransinc.com/sites/lupusqol/instrumentinformation/instrument-scoring

To compute the LupusQOL raw domain score, sum the values of the responses to each question by domain based on the tables below and divide by the number of items. Then, transform the raw domain score by dividing by 4 and multiplying by 100.

| Item<br>Respons | All the time | Most of the time | A good bit of the time | Occasionally | Never | Not applicable |
|---|---|---|---|---|---|---|
| Score | 0 | 1 | 2 | 3 | 4 | Do not score |

| Domain | Number of Items | Item Numbers |
|-----------------------|-----------------|--------------|
| Physical Health | 8 | 1-8 |
| Pain | 3 | 9-11 |
| Planning | 3 | 12-14 |
| Intimate Relationship | 2 | 15, 16 |
| Burden to Others | 3 | 17-19 |
| Emotional Health | 6 | 20-25 |
| Body Image | 5 | 36-30 |
| Fatigue | 4 | 31-34 |




## C4. Scoring algorithm for Patient Global Assessment

The Patient Global Assessment is a 10 cm visual analog scale with 0 being very well and 10 very poor. The score on this instrument is taken directly from the mark made by the patient on the VAS.



#### **Appendix D. Analytical Windows**

The last measurement for the endpoint of interest taken prior to or on the first dose of IP in this study, unless stated otherwise, will be defined as a baseline visit and the analysis visit name will be 'Baseline'. For any visit up to Day 1 pre-dose which is not a baseline visit, the analysis visit will be 'Pre-analysis'.

Since the actual visit for a subject may not exactly coincide with their scheduled visit date, to allow for variations in scheduling, the following visit windows will be used to assign evaluations to a most appropriate nominal visit for analysis and summarization. Furthermore, there will be no gaps between visit windows in order to include as many data points as possible for summarization.

If more than one actual visit (including the unscheduled visits) falls within the same defined window, the visit closest to the target day with non-missing data will be considered for analysis. If two actual visit dates are at the same distance from the target day, the latest visit with non-missing data will be considered for analysis.

The rules above for selecting a visit from multiple ones within the same visit window are not applicable to retest values of lab data. If the lab measurement is a retest, the retest value will be used.

Efficacy assessment (tender/swollen joint count, hSLEDAI, BILAG, PGA VAS, PGA 4-Point Verbal Rating Scale, CLASI), weight, and laboratory assessment (anti-dsDNA, C3 and C4 complement, chemistry, urinalysis)

| Study Visit | Target Day | Study Day |
|-------------|------------|--------------------------------------------|
| Baseline | 1 | Last evaluation prior to or on Study Day 1 |
| Week 4 | 29 | 2 - 42 |
| Week 8 | 57 | 43 - 70 |
| Week 12 | 85 | 71 - 98 |
| Week 16 | 113 | 99 - 126 |
| Week 20 | 141 | 127 - 154 |
| Week 24 | 169 | 155 - 182 |
| Week 28 | 197 | 183 - 210 |



| Week 32 | 225 | 211 - 238 |
|---------|-----|-----------|
| Week 36 | 253 | 239 - 266 |
| Week 40 | 281 | 267 - 294 |
| Week 44 | 309 | 295 - 322 |
| Week 48 | 337 | 323 - 350 |
| Week 52 | 365 | 351 - 394 |

## Hematology

| Study Visit | Target Day | Study Day |
|-------------|------------|--------------------------------------------|
| Baseline | 1 | Last evaluation prior to or on Study Day 1 |
| Week 4 | 29 | 2 - 42 |
| Week 8 | 57 | 43 - 70 |
| Week 12 | 85 | 71 - 98 |
| Week 16 | 113 | 99 - 126 |
| Week 20 | 141 | 127 - 154 |
| Week 24 | 169 | 155 - 182 |
| Week 28 | 197 | 183 - 210 |
| Week 32 | 225 | 211 - 238 |
| Week 36 | 253 | 239 - 266 |
| Week 40 | 281 | 267 - 294 |
| Week 44 | 309 | 295 - 322 |
| Week 48 | 337 | 323 - 350 |
| Week 52 | 365 | 351 - 378 |
| Week 56 | 393 | ≥ 379 |

## Vital sign

| Study Visit Target Day | Study Day |
|------------------------|-----------|
|------------------------|-----------|



| Baseline | 1 | Last evaluation prior to or on Study Day 1 |
|----------|-----|--------------------------------------------|
| Week 2 | 15 | 2 - 21 |
| Week 4 | 29 | 22 - 35 |
| Week 6 | 43 | 36 - 49 |
| Week 8 | 57 | 50 - 63 |
| Week 10 | 71 | 64 - 77 |
| Week 12 | 85 | 78 - 91 |
| Week 14 | 99 | 92 - 105 |
| Week 16 | 113 | 106 - 119 |
| Week 18 | 127 | 120 - 133 |
| Week 20 | 141 | 134 - 147 |
| Week 22 | 155 | 148 - 161 |
| Week 24 | 169 | 162 - 175 |
| Week 26 | 183 | 176 - 189 |
| Week 28 | 197 | 190 - 203 |
| Week 30 | 211 | 204 - 217 |
| Week 32 | 225 | 218 - 231 |
| Week 34 | 239 | 232 - 245 |
| Week 36 | 253 | 246 - 259 |
| Week 38 | 267 | 260 - 273 |
| Week 40 | 281 | 274 - 287 |
| Week 42 | 295 | 288 - 301 |
| Week 44 | 309 | 302 - 315 |
| Week 46 | 323 | 316 - 329 |
| Week 48 | 337 | 330 - 343 |
| Week 50 | 351 | 344 - 357 |




| Week 52 | 365 | 358 - 378 |
|---------|-----|-----------|
| Week 56 | 393 | ≥ 379 |

## Anti-phospholipid antibodies

| Study Visit | Target Day | Study Day |
|-------------|------------|--------------------------------------------|
| Baseline | 1 | Last evaluation prior to or on Study Day 1 |
| Week 24 | 169 | 2 - 266 |
| Week 52 | 365 | 267 - 378 |

## SF-36v2, PROMIS Fatigue SF 7A, LupusQoL

| Study Visit | Target Day | Study Day |
|-------------|------------|--------------------------------------------|
| Baseline | 1 | Last evaluation prior to or on Study Day 1 |
| Week 4 | 29 | 2 - 56 |
| Week 12 | 85 | 57 - 98 |
| Week 24 | 169 | 99 - 210 |
| Week 36 | 253 | 211 - 308 |
| Week 52 | 365 | 309 - 394 |





# Appendix E. Handling of Dates, Incomplete Dates and Missing Dates The reference date for the following rules is the date of first dose efavaleukin alfa.

| | | Stop Date | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Complete: yyyymmdd | | Partial:<br>yyyymm | | Partial: | | Missing |
| Start Date | | < 1 <sup>st</sup><br>dose | ≥ 1 <sup>st</sup><br>dose | < 1 <sup>st</sup><br>dose<br>yyyymm | ≥ 1 <sup>st</sup><br>dose<br><i>yyyymm</i> | < 1 <sup>st</sup><br>dose<br><i>yyyy</i> | ≥ 1 <sup>st</sup><br>dose<br><i>yyyy</i> | |
| Partial: | = 1 <sup>st</sup> dose | 2 | 1 | n/a | 1 | n/a | 1 | 1 |
| | ≠ 1 <sup>st</sup> dose | | 2 | 2 | 2 | 2 | 2 | 2 |
| Partial: | = 1 <sup>st</sup> dose | 3 | 1 | 3 | 1 | n/a | 1 | 1 |
| | ≠ 1 <sup>st</sup> dose | | 3 | | 3 | 3 | 3 | 3 |
| Missing | | 4 | 1 | 4 | 1 | 4 | 1 | 1 |

<sup>1=</sup>Impute the date of first dose or the randomization date if not treated; 2=Impute the first of the month; 3=Impute January 1 of the year; 4=Impute January 1 of the stop year

Note: For subjects who were never treated (first dose date is missing), partial start dates will be set to the first day of the partial month or first day of year if month is also missing.

#### Imputation Rules for Partial or Missing Stop Dates

Initial imputation

- If the month and year are present, impute the last day of that month.
- If only the year is present, impute December 31 of that year.
- If the stop date is entirely missing, assume the event or medication is ongoing.

If the imputed stop date is before the start date, set stop date to missing.

If the imputed stop date is after the death date, impute as death date.

